CLINICAL TRIAL: NCT02648243
Title: Impact of a Pharmacist-delivered Discharge and Follow-up Intervention for Patients With Acute Coronary Syndromes in Qatar: a Randomized Controlled Trial
Brief Title: Impact of a Pharmacist-delivered Discharge and Follow-up Intervention for Patients With Acute Coronary Syndromes in Qatar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Principal Investigator, Dr. Maguy El Hajj, Dr. Maguy El Hajj, Qatar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Qatar U
Record Dates: First submitted 2016-01-03; First posted 2016-01-07 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Coronary Syndromes
Keywords: Qatar; Acute Coronary Syndrome; Pharmacist; Medication burden; Mortality; Readmission; Adherence; Impact
MeSH Terms: conditions — Acute Coronary Syndrome; Tooth, Impacted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Patients will receive routine discharge instructions and medication information by the nurses and treating physicians at hospital discharge: Patients will not have any contact with the clinical pharmacists.
- Pharmacist delivered usual care at discharge (No Intervention): Patients will receive the usual counseling at discharge by the clinical pharmacists.
- structured intervention at discharge and tailored follow up (Experimental): The pharmacist will deliver a structured personalized discharge intervention in addition to 2 follow-up session (around 30 minutes each session) at 4 weeks of discharge and 8 weeks of discharge.
  Interventions: Behavioral: Structured intervention at discharge and tailored follow up post discharge

INTERVENTIONS:
Behavioral: Structured intervention at discharge and tailored follow up post discharge — At discharge, pharmacist-delivered personalized intervention would include the following (30-60 minutes session): The pharmacist will perform medication reconciliation and will check the appropriateness and accuracy of discharge medications. - Other potential interventions that could be done by the pharmacist include in addition to medication initiation: dose and/or frequency optimization, changing ACEI with ARB if necessary, changing to another statin if needed, identification of inappropriate or duplicated therapy, etc.
  The pharmacist will ensure that a follow-up plan for medication monitoring after discharge is communicated to the patient. The pharmacist will also provide a tailored and thorough counseling to the patient. In addition to the pharmacist delivered intervention at discharge (as described above), the study pharmacist will schedule 2 follow-up sessions (30-60 minutes each session) with the patients at 4 weeks of discharge and at 8 weeks of discharge.
  Arms: structured intervention at discharge and tailored follow up

SUMMARY:
In Qatar, cardiovascular diseases (CVD) have become the leading cause of morbidity and mortality over the past two decades. Between 1991 and 2010, a total of 16,736 patients were admitted with ACS (Acute Coronary Syndrome) in Qatar. Despite the use of percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG), and pharmacological agents to acutely reduce vascular risk, ACS patients are at high risk of having further cardiovascular events. Consequently, secondary cardiovascular risk reduction therapy is needed for all CAD (Coronary Artery Disease) patients. Clinical practice guidelines recommend that following ACS, patients should receive indefinite treatment with aspirin, a beta blocker, an angiotensin converting enzyme inhibitor (ACEI) or alternatively angiotensin II receptor blocker (ARB) and a statin. Less than 80% of ACS patients in Qatar use this quadruple combination after discharge. This creates a significant opportunity for pharmacists to improve CVD management and outcomes in Qatar. Nothing is known about the impact of Qatar clinical pharmacists as direct patient-care team members at discharge and post-discharge on the short-term and long-term outcomes of ACS patients. The proposed study is aimed to determine this impact. The investigators hypothesize that a clinical pharmacist-delivered intervention consisting of medication reconciliation and counseling at discharge and tailored follow-up post-discharge will decrease hospital readmissions, emergency department (ED) visits and all-cause mortality at 3 month, 6 months and 12 months after hospital discharge when compared with control arm and pharmacist delivered intervention at discharge only among ACS patients. The investigators also hypothesize that the effect of the intervention will increase patients' adherence to evidence-based secondary prevention medications for CAD (Coronary Artery Disease), and patient satisfaction with pharmacy services. Besides, this intervention will reduce the treatment burden on patients.

DETAILED DESCRIPTION:
Nothing is known about the impact of Qatar clinical pharmacists as direct patient-care team members at discharge and post-discharge on the short-term and long-term outcomes of patients with ACS at Heart Hospital in Qatar. This research project aims to determine this.

The investigators hypothesize that a clinical pharmacist-delivered intervention consisting of medication reconciliation and counseling at discharge and tailored follow-up post-discharge will decrease hospital readmissions, emergency department (ED) visits and all-cause mortality at 3 months, 6 months and 12 months after hospital discharge when compared with control arm and pharmacist delivered intervention at discharge only among ACS patients. The investigators also hypothesize that the effect of the intervention will increase patients' adherence to evidence-based secondary prevention medications for CAD, and patient satisfaction with pharmacy services. besides, this intervention will reduce the treatment burden on patients.

Study objectives:

1. To evaluate the effectiveness of clinical pharmacist-delivered intervention at discharge and tailored follow-up post-discharge on decreasing hospital readmissions, ED visits and mortality in ACS patients.
2. To evaluate the effectiveness of the intervention on improving patient adherence to evidence-based secondary prevention CAD medications.
3. To study the effect of the intervention on reducing the burden of treatment on patients.
4. To assess the effect of the intervention on increasing patient satisfaction with pharmacy services at Heart Hospital in Qatar.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Admitted to and discharged from any nonsurgical cardiology service at Heart Hospital with a diagnosis of ACS in the period from September 2015 to February 2016.

Exclusion Criteria:

* Severe visual impairment
* Severe hearing impairment
* Inability to communicate in English or Arabic
* Mental or psychiatric illness
* Delirium or severe dementia
* Cognitive impairment
* Incomprehensible speech
* Planned discharge to a location other than home (e.g. long-term care facility, nursing home, other medicine units etc.)
* Plan for coronary artery bypass graft (CABG) surgery during hospitalization
* Plan to leave Qatar in the next 12 months
* A terminal illness with a high likelihood of death in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
All-cause hospitalizations and cardiac-related hospital readmissions | 3 months post discharge
  This will be measured by the number (%) of hospital readmissions including hospitalizations for cardiac events, including coronary events, exacerbation of heart failure or arrhythmia. Coronary events will be defined as ACS, percutaneous coronary intervention, and/or coronary artery bypass graft. This outcome will be assessed by checking the Heart Hospital (HH) and Hamad Medical Corporation (HMC) medical records
All-cause hospitalizations and cardiac-related hospital readmissions | 6 months post discharge
  This will be measured by the number (%) of hospital readmissions including hospitalizations for cardiac events, including coronary events, exacerbation of heart failure or arrhythmia. Coronary events will be defined as ACS, percutaneous coronary intervention, and/or coronary artery bypass graft. This outcome will be assessed by checking the Heart Hospital (HH) and Hamad Medical Corporation (HMC) medical records
All-cause hospitalizations and cardiac-related hospital readmissions | 12 months post discharge
  This will be measured by the number (%) of hospital readmissions including hospitalizations for cardiac events, including coronary events, exacerbation of heart failure or arrhythmia. Coronary events will be defined as ACS, percutaneous coronary intervention, and/or coronary artery bypass graft. This outcome will be assessed by checking the Heart Hospital (HH) and Hamad Medical Corporation (HMC) medical records

SECONDARY OUTCOMES:
All-cause mortality including cardiac-related mortality | 3 months, 6 months, and 12 months post discharge
  This outcome will be measured by the number (%) of deaths. It will be assessed by checking HH and HMC medical records during the designated follow-up periods. •
ED visits including cardiac-related ED visits | 3 months, 6 months, and 12 months post discharge
  This outcome will be measured by the number (%) of ED visits. The outcome will be assessed by checking HH and HMC medical records
Patient adherence to evidence-based secondary prevention medications for CAD | 3 months, 6 months, and 12 months post discharge
  Adherence will be measured from the refill records as well as by asking the patients to list the medications they are currently taking and by using the ARMS tool
Burden of medications | 3 months, 6 months, and 12 months post discharge
  will be assessed using a questionnaire that will be adapted from a validated and translated questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Maguy El Hajj, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] El Hajj MS, Kaddoura R, Abu Yousef SEA, Orabi B, Awaisu A, AlYafei S, Shami R, Mahfoud ZR. Effectiveness of a structured pharmacist-delivered intervention for patients post-acute coronary syndromes on all-cause hospitalizations and cardiac-related hospital readmissions: a prospective quasi-experimental study. Int J Clin Pharm. 2023 Jun;45(3):630-640. doi: 10.1007/s11096-023-01538-4. Epub 2023 Feb 16. PMID 36795303
- [Derived] Zidan A, Awaisu A, Kheir N, Mahfoud Z, Kaddoura R, AlYafei S, El Hajj MS. Impact of a pharmacist-delivered discharge and follow-up intervention for patients with acute coronary syndromes in Qatar: a study protocol for a randomised controlled trial. BMJ Open. 2016 Nov 18;6(11):e012141. doi: 10.1136/bmjopen-2016-012141. PMID 27864247